CLINICAL TRIAL: NCT03692559
Title: The Effects of Different Ways of Dressing Central Line Associated Bloodstream Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, Teng,Meng-Lan Head Nurse, Head Nurse, National Taiwan University Hospital Hsin-Chu Branch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 104-032-E
Record Dates: First submitted 2017-10-18; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: CRBSI; CLABSI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- full sterile dressing (Experimental): Patients receive full sterile dressing
  Interventions: Other: full aseptic dressing
- usual standard care (No Intervention): Patients receive usual standard care

INTERVENTIONS:
Other: full aseptic dressing — Replacement of the central venous catheters in the dressing process
  Arms: full sterile dressing

SUMMARY:
The goal of our study was to investigate whether different methods of dressing could lower catheter-associated bloodstream infections.

DETAILED DESCRIPTION:
The study method was experimental in design and recruited 331 medical intensive care unit patients with placement of central catheters in one regional hospital in northern Taiwan. The investigators used block randomization to assign patients to the study group or control group. In study group which included 163 participants, the investigators used aseptic coverings during dressing and in the control group which included 168 participants the process of dressing was as routine. Study period started from the first day of catheter insertion and ends with either the removal of catheter or discharge from intensive care unit. The investigators defined the infection outcome according to culture results, and the guidelines by Infectious Diseases Society of America and Centers for Disease Control and Prevention, USA. Analysis was done by SPSS version 23. The investigators used percentage and average to study characteristics of participants. The investigators used Chi-Square or Fisher's exact test and Poisson distribution to analyze the incidence rate of bloodstream infections and the infection density. The investigators used Kaplan-Meier curve to demonstrate the catheter infection-free days and the catheter redness symptoms days of the two groups. The investigators used logistic regression model to analyze factors associated with development of bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 20 years old
* Patients with central venous catheters
* Agree to participate in this study, and fill out the study consent

Exclusion Criteria:

* PICC patients placed
* Patients with bloodstream infection
* Patients with immunocompromised patients (such as HIV, AIDS, pregnant, or cancer patients who are receiving chemotherapy or radiotherapy)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Catheter-related blood stream infections density after dressing change | up to 18 months
  Confirm blood culture results and judge whether it is catheter related Bloodstream infection(CRBSI)

SECONDARY OUTCOMES:
Central Line-Associated Bloodstream Infection density after dressing change | up to 18 months
  Confirm blood culture results and judge whether it is catheter related Bloodstream infection, CLABSI

CONTACTS AND LOCATIONS:
Overall Officials: Meng-lan Teng, Study Chair — National Taiwan University Hospital Hsin-Chu Branch

IPD SHARING:
Plan to Share IPD: No